CLINICAL TRIAL: NCT06743646
Title: A Multicenter, Randomized，Controlled，Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of ZVS101e Administered as a Single Subretinal Injection in Subjects With Bietti's Crystalline Dystrophy (BCD)
Brief Title: Efficacy and Safety of ZVS101e in Patients With Bietti 's Crystalline Dystrophy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chigenovo Co., Ltd (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZYA-2024-001
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Bietti Crystalline Corneoretinal Dystrophy; Bietti Crystalline Dystrophy
Keywords: gene replacement therapy; ZVS101e; AAV8-hCYP4V2; phase 3; Bietti crystalline corneoretinal dystrophy
MeSH Terms: conditions — Bietti Crystalline Dystrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): Each Participant in this group will receive a unilateral subretinal injection of ZVS101e in the study eye
  Interventions: Drug: ZVS101e
- Control group (No Intervention): Participants in the control group will receive no treatment

INTERVENTIONS:
Drug: ZVS101e — subretinal injection of ZVS101e
  Other Names: AAV8-hCYP4V2; AAV2/8-hCYP4V2; Puliretgene parvec
  Arms: Treatment group

SUMMARY:
This is a multi-center, randomized and controlled phase 3 clinical trial.

DETAILED DESCRIPTION:
Subjects who have signed the written informed consent form and who were eligible for enrollment after screening will be randomly assigned to the treatment group or untreated control group. Each Participant in the treatment group will receive a unilateral subretinal injection of ZVS101e in the study eye.

Participants in the control group will receive no treatment during the first 52 weeks of enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. All of the following inclusion criteria should be met for enrollment into the trial:
2. Fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial and sign the informed consent form, and be able to complete all trial procedures as required by the protocol;
3. Clinical diagnosis of Bietti's crystalline dystrophy (BCD), age≥18 years ;
4. Genetic testing confirmed biallelic CYP4V2 mutations without other ophthalmic genetic diseases;
5. Best-corrected visual acuity of 5-60 ETDRS letters.

Exclusion Criteria:

1. The study eye has or has had macular lesions such as macular hole or macular neovascularization; glaucoma, diabetic retinopathy, or any other ocular disease that may preclude surgery or interfere with interpretation of the study endpoints
2. The study eye had received the following intraocular surgical treatments: retinal reattachment, vitrectomy;
3. The study eye had received any intraocular surgery, such as phacoemulsification 3 months prior to enrollment;
4. Previously treatment of either eye with gene therapy or stem cell therapy for BCD and other ocular diseases, including but not limited to viral vector gene therapy, RNA therapy;
5. Pregnant or lactating women;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of study eyes with a ≥15-letter improvement from baseline in BCVA | From baseline to Week 52
  Best corrected visual acuity (BCVA) will be assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart. A 15-letter improvement over the baseline is clinical meaningful.

SECONDARY OUTCOMES:
Change from Baseline in BCVA | From baseline to Week 52
  Best corrected visual acuity (BCVA) will be assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart. The larger the letter number, the better the vision.
Proportion of study eyes with a ≥10-letter improvement from baseline in BCVA | From baseline to Week 52
  Best corrected visual acuity (BCVA) will be assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart.
Change from baseline in multi-luminance mobility test (MLMT) score | From baseline to Week 52
  MLMT will be assessed using both eyes at different levels of illumination. A higher score indicates better functional vision.
Change from baseline in 25-Item visual function questionnaire (VFQ-25) score | From baseline to Week 52
  National eye institute 25-item visual function questionnaire (NEI VFQ-25) consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively.
Change from Baseline in microperimetry | From baseline to Week 52
  Microperimetry will be measured using MP-3，changes in retinal sensitivity (dB) will be analyzed.
Change from baseline in OCT | From baseline to Week 52
  Retinal thickness will be assessed using OCT.
Incidence and severity of ocular and systemic adverse events | From baseline to Week 52
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event will not need to have a causal relationship with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jinlu Zhang, MD, Study Director — Chigenovo Co., Ltd
Locations (8):
- China (8):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality
  - Eye Hospital, Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jia R, Meng X, Chen S, Zhang F, Du J, Liu X, Yang L. AAV-mediated gene-replacement therapy restores viability of BCD patient iPSC derived RPE cells and vision of Cyp4v3 knockout mice. Hum Mol Genet. 2023 Jan 1;32(1):122-138. doi: 10.1093/hmg/ddac181. PMID 35925866
- [Result] Wang J, Zhang J, Yu S, Li H, Chen S, Luo J, Wang H, Guan Y, Zhang H, Yin S, Wang H, Li H, Liu J, Zhu J, Yang Q, Sha Y, Zhang C, Yang Y, Yang X, Zhang X, Zhao X, Wang L, Yang L, Wei W. Gene replacement therapy in Bietti crystalline corneoretinal dystrophy: an open-label, single-arm, exploratory trial. Signal Transduct Target Ther. 2024 Apr 24;9(1):95. doi: 10.1038/s41392-024-01806-3. PMID 38653979